CLINICAL TRIAL: NCT06979947
Title: Effect of Structured Education on Menopause-Specific Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Tuba Enise BENLI, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Record Dates: First submitted 2025-05-10; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Menopause; Quality of Life
Keywords: Menopause; Structured Education; Midwifery; MENQOL; Women's Health

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either an intervention group receiving structured education or a control group receiving no intervention.
Masking Description: The study was not blinded; both participants and investigators were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants received a structured menopause education program delivered by a midwife. The program consisted of four weekly sessions, each lasting 20-25 minutes, covering menopause-related symptoms, physiological changes, and coping strategies. Educational materials were developed by the researchers and validated by experts. The education was tailored based on participants' MENQOL pre-test scores.
  Interventions: Behavioral: Structured Menopause Education Program
- Control Group (No Intervention): Participants received no intervention during the study. They completed the same assessments at the same time points as the intervention group. After final data collection, the educational material was shared with them to ensure equity.

INTERVENTIONS:
Behavioral: Structured Menopause Education Program — The structured education program was developed by midwifery researchers and delivered face-to-face by a certified midwife over four weekly sessions. Each session lasted approximately 20-25 minutes and covered topics such as menopausal symptoms, lifestyle changes, and coping strategies. Educational materials were individualized based on participants' MENQOL pre-test scores.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the impact of a structured education program delivered under midwife guidance on menopause-specific quality of life among women aged 45-55 undergoing natural menopause, and to assess the sustainability of its effects over time.

DETAILED DESCRIPTION:
This randomized controlled longitudinal study was conducted with 101 women aged 45-55 experiencing natural menopause (intervention: 51, control: 50). The intervention group received a structured menopause education program developed based on literature and expert review. Data were collected using a Personal Information Form and the Menopause-Specific Quality of Life Questionnaire (MENQOL) at three time points: baseline (T1), after education (T2), and six months later (T3). The intervention consisted of four weekly face-to-face sessions delivered by a midwife. The education content included information on menopausal changes, symptoms, and coping strategies. The control group received no intervention during the study but received educational material after final data collection. Data were analyzed using SPSS 20.0 with p<0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 45-55

  * Experiencing natural (non-surgical) menopause
  * Literate and able to complete questionnaires
  * No neurological or cognitive impairments
  * Willing to participate and attend sessions
  * Has access to phone/internet

Exclusion Criteria:

* Surgical menopause
* Hormonal disorders causing amenorrhea
* Current use of hormonal therapy or antidepressants
* Diagnosed psychiatric conditions

Removal Criteria (if applicable):

* Did not attend at least 80% of sessions
* Lost to follow-up at 6 months
* Developed a new health issue affecting menopause
* Participated in other menopause interventions
* Incomplete or inconsistent questionnaire

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Menopause-Specific Quality of Life (MENQOL) Scores | Baseline (T1), 4 weeks after intervention (T2), and 6 months after intervention (T3)
  Mean change in total and subscale scores of the Menopause-Specific Quality of Life Questionnaire (MENQOL) from baseline to 6-month follow-up. Higher scores indicate greater symptom severity and lower quality of life.The MENQOL total score ranges from 0 to 6. Higher scores indicate greater symptom severity and lower quality of life.

SECONDARY OUTCOMES:
Change in MENQOL Subscale Scores (Vasomotor, Psychosocial, Physical, Sexual) | Baseline, 4 weeks, and 6 months
  Comparison of MENQOL subscale scores between intervention and control groups at each time point. Subscales include vasomotor, psychosocial, physical, and sexual symptoms.Each MENQOL subscale (vasomotor, psychosocial, physical, sexual) has items scored from 0 to 6. Higher scores reflect more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: KADER ATABEY, Principal Investigator — Inonu University
Locations (1):
- Hasköy Family Health Center, Muş, CİTY, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD).